CLINICAL TRIAL: NCT07114640
Title: Far Eastern Memorial Hospital
Brief Title: The Effect of Nighttime Mirabegron, Solifenacin, Tolterodine, or Oxybutynin on Nocturia, Sexual Function, Autonomic Function, and Lower Urinary Tract Blood Flow Perfusion in Women With Overactive Bladder Syndrome: Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief and Professor, Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110416-F
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Urinary Bladder, Overactive
Keywords: autonomic nerve system, nocturia, psychologic distress, sexual function, bladder blood perfusion, heart rate variability, overactive bladder syndrome
MeSH Terms: conditions — Urinary Bladder, Overactive; Nocturia | interventions — mirabegron; Solifenacin Succinate; Tolterodine Tartrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- mirabegron (Active Comparator): mirabegron 25 mg
  Interventions: Drug: Mirabegron 25mg
- Solifenacin (Active Comparator): Solifenacin 5mg
  Interventions: Drug: Solifenacin 5 mg
- Tolterodine (Active Comparator): Tolterodine 4mg
  Interventions: Drug: Tolterodine 4 mg
- Oxybutynin ER (Active Comparator): Oxybutynin ER 5mg
  Interventions: Drug: Oxybutynin ER 5 mg

INTERVENTIONS:
Drug: Mirabegron 25mg — Taking 25 mg mirabegron in the nighttime
  Arms: mirabegron
Drug: Solifenacin 5 mg — Taking 5 mg solifenacin in the nighttime
  Arms: Solifenacin
Drug: Tolterodine 4 mg — Taking 5 mg tolterodine in the nighttime
  Arms: Tolterodine
Drug: Oxybutynin ER 5 mg — Taking 5 mg oxybutynin ER in the nighttime
  Arms: Oxybutynin ER

SUMMARY:
The optimal medication for women with nocturia remains uncertain. This clinical trial aimed to determine the most effective medication for women with overactive bladder and nocturia. Its primary objectives were to answer the following questions:

Which medication is most effective for women with nocturia? Which medication has the least effect on heart rate variability in women with nocturia?

DETAILED DESCRIPTION:
We will conduct a prospective randomized controlled study in the outpatient clinic of Department of Obstetrics and Gynecology of Far Eastern Memorial Hospital. All female patients with overactive bladder syndrome enrolled in the study will be requested to fill in the questionnaires and before taking the drug and four weeks and twelve weeks after taking the medication. In addition, measurement of heart rate variability will be performed before and twelve weeks after taking the medication. All enrolled women will be randomized to receive nighttime mirabegron, solifenacin, tolterodine or oxybutynin for 12 weeks.

The aims of this study is to obtain the impact of nighttime dosing of mirabegron, solifenacin, tolterodine or oxybutynin versus combined therapy on nocturia, psychologic distress, sexual function, cognition, heart rate variability and bladder blood perfusion in women with overactive bladder syndrome.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old.
* female patients with overactive bladder syndrome

Exclusion Criteria:

* Clinically significant dysuria (inability to urinate, difficulty urinating).
* Severe stress urinary incontinence (urinary incontinence caused by coughing).
* Mixed urinary incontinence mainly caused by stress urinary incontinence (urinary incontinence caused by coughing as the main symptom).
* Contraindications to antimuscarinic drugs or adrenergic receptor agonists.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-08-07 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Improvement of overactive bladder symptoms | 12 weeks
  Comparisons of the changes of overactive bladder symptom score between groups

SECONDARY OUTCOMES:
Change of heart rate variability | 12 weeks
  Comparisons of the changes of heart rate variability between groups
Change of bladder blood perfusion | 12 weeks
  Comparisons of the changes of bladder blood perfusion between groups

OTHER OUTCOMES:
Change of quality of life | 12 weeks
  Comparisons of the change of King's Health Questionnaire score between groups

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital,, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No